CLINICAL TRIAL: NCT02384499
Title: Treatment of Fecal Incontinence Using Allogenic-Adipose-derived Mesenchymal Stem Cells: A Prospective, Dose Escalation, Randomized, Placebo-controlled, Parallel-group, Single-blind, Single-center Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2014-0271
Record Dates: First submitted 2015-02-24; First posted 2015-03-10 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Saline Solution; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALLO-ASC group (Experimental): Allogenic-adipose-derived mesenchymal stem cell (ALLO-ASC) with fibrin glue injection to the anal sphincter
  Interventions: Biological: ALLO-ASC injection
- Normal saline group (Placebo Comparator): 0.9% normal saline with fibrin glue injection to the anal sphincter
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ALLO-ASC injection — Allogenic-adipose-derived mesenchymal stem cells (ALLO-ASC) injection to the anal sphincter of patients with fecal incontinence
  Other Names: ALLO-ASC
  Arms: ALLO-ASC group
Drug: Placebo — 0.9% normal saline with fibrin glue injection to the anal sphincter of patients with fecal incontinence
  Other Names: Normal saline with fibrin glue injection
  Arms: Normal saline group

SUMMARY:
* Purpose: The investigators aimed to investigate the safety and efficacy in the treatment of fecal incontinence by injection of ALLO-ASC into the anal sphincter.
* Method

  1. Safety test of allogenic ASCs injection
  2. Efficacy test of allogenic ASCs injection

DETAILED DESCRIPTION:
* Background: Fecal incontinence is a distressing condition with recurrent uncontrolled passage of fecal material. Although fecal incontinence is developed by multifactorial causes, treatments were limited in medical or surgical methods. According to the recent studies of stem cell regeneration, it is reported that human adipose-derived stem cells have plentiful capacity in muscle regeneration, which had the efficacy to treat Crohn's fistulas. Therefore, the investigators hypothesized that the capability of muscle regeneration of allogenic-adipose-derived mesenchymal stem cells (ALLO-ASC) can be used to treat degenerated anal sphincter, which leads to fecal incontinence.
* Purpose:The investigators aimed to investigate the safety and efficacy in the treatment of fecal incontinence by injection of ALLO-ASC into the anal sphincter.
* Method

  1. Safety test of allogenic ASCs injection In the first year, the investigators will investigate the safety of ALLO-ASC injection by a dose escalation study. Patients are sequentially enrolled into three groups, which are composed of three patients each. They are treated with an injection of ALLO-ASC to the anal sphincter for 3x107 cells/ml (group 1), 6x107 cells/ml (group 2), 9x107 cells/ml (group 3), respectively. After receiving the ALLO-ASC injection, patients will receive a physical examination, a serologic and immunologic response test (CD4/CD8) with an assessment of the Wexner score, patient satisfaction survey, WHO toxicity scale, adverse events, anorectal manometry and endorectal ultrasound at 1, 4, 8 weeks, 4, 6, 9, and 12 months in the outpatient clinic. The response of ALLO-ASC injection is assessed at 8 weeks after an injection and the most effective dose is determined among the groups.
  2. Efficacy test of allogenic ASCs injection In the second year, the investigators will assess the efficacy of the ALLO-ASC injection comparing the ALLO-ASC injection group and the placebo group (0.9% normal saline injection) by a randomized, open-label, single-blind design. Each group is composed of six patients. Both the clinical assessment and follow-up period are identical with the first-year protocol.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years old
* Patients who received either medical therapy or biofeedback for fecal incontinence for more than 2 months with Wexner score ≥ 8
* Transanal ultrasonography: presents a continuous fashion of anal sphincter
* Anal manometery: decreased anal pressures than normal level
* Negative for urine β-hCG in the screening test
* An informed consent form has been signed by the patient

Exclusion Criteria:

* Participation in another clinical trial within 30 days
* History of anorectal surgery within the previous 6 months
* History of malignant tumor surgery within the previous 5 years (except for carcinoma in situ)
* Patients requiring anorectal surgical treatments
* History of artificial sphincter surgery
* History of vaginal delivery within 6 months
* Medical history of variant Creutzfeld-Jakobs disease or related diseases
* Allergy to bovine-derived materials, fibrin glue or anesthestics
* Autoimmune disease
* Active tuberculosis
* Pregnant or breastfeeding women
* Unwillingness to use contraceptive methods
* Patients with inflammatory bowel disease
* Alcohol or drug-abuse
* Use of cytotoxic agents within 30 days
* Patients who have severe constipation (<2 times/week), anal fistula, rectal prolapse, spinal cord injury, multiple sclerosis, Parkinson's disease
* Patients with one of hematologic disease, immunodeficieny, fever, acute disease or severe chronic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Clinically measured abnormality of laboratory tests and adverse events | one year (12 months)
  The investigators will assess the safety of allogenic-adipose-derived mesenchymal stem cell (ALLO-ASC) injection to the anal sphincter among the three experimental groups (group 1: 3x107 cells/ml; group 2: 6x107 cells/ml; group 3: 9x107 cells/ml)).

SECONDARY OUTCOMES:
Satisfaction as measured by Wexner Score | one year (12 months)
  Improvement of Wexner Score at 12 months compared to baseline per each group. (The investigators will assess the efficacy of the ALLO-ASC injection comparing the ALLO-ASC injection group and the placebo group (0.9% normal saline injection) by a randomized, open-label, single-blind design.)

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Colon and Rectal Surger, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] White AB, Keller PW, Acevedo JF, Word RA, Wai CY. Effect of myogenic stem cells on contractile properties of the repaired and unrepaired transected external anal sphincter in an animal model. Obstet Gynecol. 2010 Apr;115(4):815-823. doi: 10.1097/AOG.0b013e3181d56cc5. PMID 20308844
- [Background] Parmar N, Kumar L, Emmanuel A, Day RM. Prospective regenerative medicine therapies for obstetric trauma-induced fecal incontinence. Regen Med. 2014;9(6):831-40. doi: 10.2217/rme.14.56. PMID 25431918
- [Background] Kang SB, Lee HN, Lee JY, Park JS, Lee HS, Lee JY. Sphincter contractility after muscle-derived stem cells autograft into the cryoinjured anal sphincters of rats. Dis Colon Rectum. 2008 Sep;51(9):1367-73. doi: 10.1007/s10350-008-9360-y. Epub 2008 Jun 7. PMID 18536965
- [Background] Lorenzi B, Pessina F, Lorenzoni P, Urbani S, Vernillo R, Sgaragli G, Gerli R, Mazzanti B, Bosi A, Saccardi R, Lorenzi M. Treatment of experimental injury of anal sphincters with primary surgical repair and injection of bone marrow-derived mesenchymal stem cells. Dis Colon Rectum. 2008 Apr;51(4):411-20. doi: 10.1007/s10350-007-9153-8. Epub 2008 Jan 26. PMID 18224375
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Derived] Park EJ, Kang J, Baik SH. Treatment of faecal incontinence using allogeneic-adipose-derived mesenchymal stem cells: a study protocol for a pilot randomised controlled trial. BMJ Open. 2016 Feb 17;6(2):e010450. doi: 10.1136/bmjopen-2015-010450. PMID 26888731